CLINICAL TRIAL: NCT00287118
Title: A Multicentre, Open Label Phase IIIb/IV Study of Subcutaneously Administered Raptiva in the Treatment of Adult Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25161; CONTROL I Study
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2017-08

CONDITIONS: Candidates for Systemic Therapy for Psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

ARMS (1):
- Efalizumab (Experimental)
  Interventions: Drug: Efalizumab

INTERVENTIONS:
Drug: Efalizumab — Subjects will receive a conditioning dose of 0.7 milligram per kilogram (mg/kg) efalizumab subcutaneously on study Day 0 followed by 1.0 mg/kg efalizumab subcutaneously once a week for 23 weeks.
  Other Names: Raptiva

SUMMARY:
An open-label, multi-center study to establish psoriasis control of moderate to severe plaque psoriasis with Raptiva therapy administered subcutaneously for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A) In the opinion of the investigator, candidate for systemic therapy for psoriasis could include:
* Patients with moderate to severe plaque psoriasis defined by Psoriasis Area and Severity Index (PASI) less than (>) 10 and body surface area (BSA) greater than (>) 10
* Patients with the following may also be deemed to require systemic therapy in the judgement of the physician:
* Severe psychosocial disability (in the judgement of the physician), or
* Nail psoriasis, or
* Scalp psoriasis, or
* Palmar plantar psoriasis etc OR
* B) Subjects who have completed the CLEAR study investigational medicinal product (IMP) 24011 (NCT00256139) and who wish to continue Raptiva (efalizumab) therapy.
* Body weight of 120 kg
* 18 to 75 years old
* For women of childbearing potential and for men whose partner can become pregnant, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study up to 3 months after the last dose of Raptiva
* Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other ultraviolet (UV) light sources during the study
* Agreement to participate in the study
* Signed informed consent
* Discontinuation of any systemic psoriasis treatment prior to commencement of the study drug. No washout period is required for these agents prior to starting study and receiving first dose of study drug (Raptiva)
* Discontinuation of all biologic agents (other than Raptiva) 3 months prior to receiving first dose of study drug (Raptiva)
* Discontinuation of Psoralen-ultraviolet light A (PUVA), Ultraviolet light B (UVB) treatment 28 days prior to commencement of receiving first dose of study drug.
* Discontinuation of any investigational drug or treatment 3 months prior to study Day 0 or as per washout requirements from previous protocol
* No vaccinations (e.g., tetanus, booster, influenza vaccine) at least 14 days prior to first dose of study drug
* Treatment regimens of b-blockers, Angiotensin-converting enzyme (ACE) inhibitors, antimalarial drugs, quinidine, interferon, or lithium stable for at least 28 days prior to first dose of study drug

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* Active rebound of psoriasis during or following discontinuation of the previous Raptiva treatment( PASI >125% from baseline and/or new predominant morphology of psoriasis) when reason was adverse event or lack of efficacy of Raptiva. If it was due to another non drug reason (vaccination, or infection) then the patient can be included in this study.
* History of severe allergic or anaphylactic reactions to humanised monoclonal antibodies
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for human immunodeficiency virus (HIV). Patients will undergo mandatory testing at screening. Patients who are positive for HIV will be excluded.
* Pregnancy or lactation
* White blood cell (WBC) count <4000 per Liter (L) or >14,000/L
* Patient with a history of clinically significant thrombocytopenia, bleeding disorders or a platelet count < 00,000 cells/L
* Seropositivity for hepatitis B or C virus Patients will undergo testing at screening. Patients who are positive for hepatitis B antigen or hepatitis C antibody will be excluded.
* Hepatic enzymes >3 times the upper limit of normal
* History of active tuberculosis (TB) or currently undergoing treatment for TB within one year prior to study Day 0. Chest X-ray (within 3 months prior to Study Day 0) is required for high-risk patients. Patients with a positive chest X-ray will be excluded.
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders. Patients with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled.
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Serum creatinine >2 times the upper limit of normal
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
* History of substance abuse within the last 5 years
* Any medical condition that, in the judgment of the investigator, would jeopardize the patient's safety following exposure to study drug

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2004-10-27 (Actual); Primary Completion 2006-05-30 (Actual); Study Completion 2006-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Medical Information Switzerland, Geneva, Switzerland

REFERENCES:
- [Result] Stengel FM, Petri V, Campbell GA, Dorantes GL, Lopez M, Galimberti RL, Valdez RP, de Arruda LF, Guerra MA, Chouela EN, Licu D; International IMP25161 Study Group. Control of Moderate-to-Severe Plaque Psoriasis with Efalizumab: 24-Week, Open-Label, Phase IIIb/IV Latin American Study Results. Arch Drug Inf. 2009 Dec;2(4):71-78. doi: 10.1111/j.1753-5174.2009.00024.x. PMID 20098510

RESULTS

PARTICIPANT FLOW:
Groups:
- Efalizumab: Subjects received a conditioning dose of 0.7 milligram per kilogram (mg/kg) efalizumab subcutaneously on study Day 0 followed by 1.0 mg/kg efalizumab subcutaneously once a week for 23 weeks.
Period: Overall Study
Arm/Group | Efalizumab
Started | 189
Completed | 137
Not Completed | 52
Not completed — Adverse Event | 30
Not completed — Death | 1
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | Efalizumab
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 134

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Physician's Global Assessment (PGA) Ratings of "Excellent" or "Cleared" at Week 24
Description: The PGA rating was used to assess the global response of all psoriatic lesions by comparing subject's present condition to baseline photographs or body diagrams. The response was classified as Cleared: 100% improvement of all clinical signs and symptoms compared to baseline; Excellent: 75% to 99% improvement of all signs and symptoms compared to baseline; Good: 50% to 74% improvement of signs and symptoms compared to baseline; Fair: 25% to 49% improvement of signs and symptoms compared to baseline; Slight: 1% to 24% improvement of signs and symptoms compared to baseline; Unchanged: Clinical signs and symptoms unchanged from baseline and Worse: Clinical signs and symptoms deteriorated from baseline.
Time Frame: Week 24
Population: The Intent to Treat (ITT) population consisted of all subjects who received at least 1 dose of trial medication.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Efalizumab
Number analyzed (Participants) | 189
percentage of subjects | 46.0 [38.9 to 53.1]

ADVERSE EVENTS:
Arm/Group | Efalizumab
Serious Adverse Events (participants affected / at risk) | 21/189
Other Adverse Events (participants affected / at risk) | 161/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=189)
Psoriasis (Skin and subcutaneous tissue disorders) | 7
Nail psoriasis (Skin and subcutaneous tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Hepatic enzyme increased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Lumbar puncture headache (Injury, poisoning and procedural complications) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab (N=189)
Headache (Nervous system disorders) | 68
Dizziness (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 2
Burning sensation (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Influenza like illness (General disorders) | 22
Pyrexia (General disorders) | 21
Chills (General disorders) | 18
Feeling hot (General disorders) | 6
Oedema peripheral (General disorders) | 6
Chest pain (General disorders) | 4
Asthenia (General disorders) | 3
Fatigue (General disorders) | 3
Malaise (General disorders) | 2
Oedema (General disorders) | 2
Pain (General disorders) | 2
Feeling cold (General disorders) | 1
Hyperthermia (General disorders) | 1
Injection site irritation (General disorders) | 1
Injection site pain (General disorders) | 1
Prostration (General disorders) | 1
Thirst (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 17
Arthritis (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Monarthritis (Musculoskeletal and connective tissue disorders) | 3
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Influenza (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 6
Herpes simplex (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Onychomycosis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Acarodermatitis (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Condyloma acuminatum (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dental caries (Infections and infestations) | 1
Dermatophytosis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Nail candida (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 11
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 6
Eosinophilia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Lymphocytosis (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1
Blood creatine phosphokinase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Culture throat positive (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Weight decreased (Investigations) | 1
Hypertension (Vascular disorders) | 9
Peripheral occlusive disease (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Conjunctivitis (Eye disorders) | 2
Eye pain (Eye disorders) | 2
Blepharitis (Eye disorders) | 1
Blepharospasm (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Growth of eyelashes (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Ear pain (Ear and labyrinth disorders) | 4
Deafness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Genital discharge (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Peyronie's disease (Reproductive system and breast disorders) | 1
Vaginal disorder (Reproductive system and breast disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Stress (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Leukocyturia (Renal and urinary disorders) | 1
Nephritis (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other